CLINICAL TRIAL: NCT06213337
Title: Evaluation of the Effectiveness of Virtual Classroom Training and SMS Supported Interventions in Improving Foot Care Behaviors and Foot Care Self-Efficacy of Diabetic Patients
Brief Title: Virtual Classroom Training and SMS Supported Interventions Improving Foot Care and Self-Efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Burak Arslan, Lecturer, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BArslan
Record Dates: First submitted 2023-12-14; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetic foot; virtual systems; Short Message Service
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (No Intervention): No intervention will be applied to this group.
- virtual classroom group (Experimental): Participants in this group will be given virtual classroom training on foot care.
  Interventions: Other: Foot care training with virtual classroom
- SMS support group (Experimental): Information regarding foot care will be sent via SMS to the participants in this group.
  Interventions: Other: Foot care training with SMS support
- SMS supported virtual classroom training group (Experimental): Participants in this group will be given virtual classroom training with SMS support.
  Interventions: Other: Foot care training with virtual classroom and SMS support

INTERVENTIONS:
Other: Foot care training with virtual classroom — Providing foot care training once every two weeks in virtual classes created via the Google meet application.
  Arms: virtual classroom group
Other: Foot care training with SMS support — Total of 60 SMS messages containing foot care information will be sent, one every day.
  Arms: SMS support group
Other: Foot care training with virtual classroom and SMS support — Providing foot care training once every two weeks in virtual classes created via the Google meet application. Furthermore, total of 60 SMS messages containing foot care information will be sent, one every day.
  Arms: SMS supported virtual classroom training group

SUMMARY:
The type of this research is a randomized controlled experimental study. The aim of the research is to determine the effectiveness of virtual classroom training and SMS support in improving foot care behaviour and foot care self-efficacy in diabetic patients.

The basic questions the research aims to answer are:

* Is virtual classroom training effective in improving foot care behaviour and foot care self-efficacy in diabetic patients?
* Are SMS-supported interventions effective in improving foot care behaviour and foot care self-efficacy in diabetic patients? Within the scope of the research, participants are expected to attend virtual classroom training and read the SMS sentences sent.

In order to examine the effects of virtual classroom training and SMS-supported interventions, researchers created a control group, a virtual classroom, an SMS support group, and an SMS-supported virtual classroom group.

ELIGIBILITY:
Inclusion Criteria:

* Reporting that you have internet, computer/smartphone access
* Becoming literate
* Ability to use the internet and mobile devices effectively
* Declaring that you are competent to use technology-based training
* Being between the ages of 18-55
* Diagnosis period of 1 year or more

Exclusion Criteria:

* Having a psychiatric/neurological disability that may prevent participation in the research
* Having any diagnosis of learning disability
* Having an existing foot ulcer
* Having a history of foot ulcers and amputation in the past
* Having severe vision problems/retinopathy
* Having severe hearing impairment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Development of foot care behavior in diabetic patients | within 3 months
  Foot Care Behavior Scale Total Score increasing
Development of foot care self-efficacy in diabetic patients | within 1 months
  Foot Care Self-Efficacy Scale Total Score increasing

CONTACTS AND LOCATIONS:
Overall Officials: Burak Arslan, Lecturer, Principal Investigator — Hitit University; Afitap Özdelikara, Assoc. Prof., Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No